CLINICAL TRIAL: NCT01285258
Title: Study of Peripartum Hysterectomy for Maternal Hemorrhage
Brief Title: Emergency Peripartum Hysterectomy: A Prospective Study in Iran
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-13
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2004-03

CONDITIONS: Postpartum Hemorrhage
Keywords: Peripartum; hysterectomy; placenta accreta; mortality
MeSH Terms: conditions — Postpartum Hemorrhage; Placenta Accreta | interventions — Hysterectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peripartum (Other): patients whom underwent peripartum hysterectomy
  Interventions: Procedure: hysterectomy

INTERVENTIONS:
Procedure: hysterectomy — excluding the uterus with saving ovaries

SUMMARY:
The purpose of this study is to determine the effects of peripartum hysterectomy for maternal hemorrhage.

DETAILED DESCRIPTION:
Emergency peripartum hysterectomy is a life-saving surgical procedure which performed to control massive hemorrhage. This study was conducted to determine the factors leading to and maternal mortality and morbidity rates among the women whose underwent peripartum hysterectomy with the focus on referral or non-referral patient status.

ELIGIBILITY:
Inclusion Criteria:

* Women who have nonresponse hemorrhage after delivery

Exclusion Criteria:

* Women who delivered before 24 weeks

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
death rate | at 2 minutes after operation

SECONDARY OUTCOMES:
urological complication | at 2 minutes after operation

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Principal Investigator — MD,research comittee
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran